CLINICAL TRIAL: NCT04032067
Title: A Randomized, Active-Controlled, Double-Blind, Parallel Design, Multi-Center, Phase III Clinical Trial to Evaluate the Efficacy and Safety of GV1001 in Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: Evaluate the Efficacy and Safety of GV1001 in Patients With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KG8/2019
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign Prostatic Hyperplasia; GV1001
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Saline Solution; Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): GV1001-Placebo ID injection administered every 2 weeks through Week 24
  + Proscar PO administered once a day through Week 24
  Interventions: Drug: GV1001 placebo
- Study Group 1 (Experimental): GV1001 0.56 mg ID injection administered every 2 weeks through Week 24
  + Proscar-placebo PO administered once a day through Week 24
  Interventions: Drug: Proscar placebo
- Study Group 2 (Experimental): GV1001 1.12 mg ID injection administered every 2 weeks through Week 24
  + Proscar-placebo PO administered once a day through Week 24
  Interventions: Drug: Proscar placebo

INTERVENTIONS:
Drug: GV1001 placebo — 0.9 % Normal Saline
  Other Names: Normal Saline
  Arms: Control Group
Drug: Proscar placebo — PO
  Other Names: Finasteride
  Arms: Study Group 1; Study Group 2

SUMMARY:
The current study is being conducted by the Sponsor to evaluate the efficacy and safety of GV1001 (0.56 mg and 1.12 mg) administered as a treatment for Benign prostate hyperplasia(BPH). The investigational drug, GV1001, was first developed as a cancer vaccine for use as active immunotherapy of cancer forms expressing telomerase (eg, pancreatic cancer, prostate cancer, etc.). Subsequently, it was found that GV1001 showed efficacy in alleviating BPH symptoms during in vivo studies by reducing the size of the prostate gland. Based on the result, the effectiveness of GV1001 as a treatment for BPH has been assessed in experimental animals that are designed to develop BPH.

It is considered that GV1001 acts to alleviate BPH and the results obtained from previous phase II study indicate that GV1001 may provide potential beneficial effects in BPH patients.

So this study is to verify the efficacy and safety of GV1001 on BPH population, large-scale clinical study than phase II.

DETAILED DESCRIPTION:
This was a multi-center, randomized, Double-blind, Active-controlled, parallel design, Phase 3 study in patients with BPH. The study consisted of a Screening period, a 4-weeks Run-in/Washout period, a 24-week Treatment period, an Evaluation and Close-out Visit at Week 24.

There are a total of 3 groups in this study, which contained 2 study groups (GV1001) and 1 placebo group (0.9% normal saline). Approximately 417 patients are planned to be randomly assigned into the study in a 1:1:1 ratio. All patients are randomized into 1 of 3 treatment groups to ensure completion of patients.

The Screening period have a time period of 4 weeks before the beginning of Run-in/Washout period. Eligible patients entered into a 4-week Run-in/Washout period and receive placebo treatment, which will be completed before randomization on Week 0. All randomized patients will receive the investigational drug or a placebo via intradermal injection 12 times with a 2-week interval at Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24. Efficacy evaluation will be conducted at Weeks 4, 8, 12, 16, 20 and 24, and safety evaluation will be conducted throughout the 24-weeks period.

ELIGIBILITY:
Inclusion Criteria:

1. A male at 50 years of age and older
2. Clinical signs and symptoms of benign prostatic hyperplasia

   1. A volume of prostate gland (TRUS) > 30 cc
   2. Moderate to severe lower urinary tract symptoms with IPSS ≥ 13
   3. 5-15 mL/sec of maximum flow rate (Qmax) measured when urine volume was at least 125 mL
3. PSA level < 10 ng/mL (however, if 4 ng/mL < PSA < 10 ng/mL, a person with a biopsy result, confirming that he does not have prostate cancer)
4. Residual urine volume ≤ 200 Ml
5. Consent not to participate in other clinical trials as a subject during this clinical trial period.
6. Consent of patient and patient's partner a. Patient

   * Consent to avoid pregnancy by using condoms for 90 days after the end of study participation period and treatment. (Not applied if the patient had vasectomy.) b. Patient's partner (Consent should be obtained before visit 4, when necessary.)
   * Consent to avoid pregnancy by using contraceptive devices or oral contraceptives during the patient's participation in clinical trial and for 90 days after the end of treatment, except if the partner reaches menopause or is surgically sterilized.

Exclusion Criteria:

1. Hypersensitivity reactions to ingredients of this drug.
2. Taking drugs that affect the results of clinical trials. ex) 5-alpha reductase inhibitors, drugs similar to LHRH, alpha blockers, alpha-beta blockers, anticholinergics, antidiuretic hormones, diuretics, PDE-5 inhibitors, beta-3 adrenoceptor antagonists, steroids, immune suppressants, saw palmetto, etc.
3. Taking drugs of an unapproved study drug in the past or the study drug for this clinical trial
4. Diagnosis with prostate cancer in the past or at present
5. Diagnosis by an investigator to have an influence to an evaluation on urine flow symptoms due to other previous or current diseases besides benign prostatic hyperplasia
6. Surgeries or radiation therapies for prostate gland, bladder or pelvis, or who had invasive treatments for benign prostatic hyperplasia
7. Severe medical condition which may be cause problem to conduct the clinical trial (e.g., chronic heart failure (CHF), difficult-to-control diabetes (HbA1c > 7%), mental disorder, drug, or alcohol abuse, etc.)
8. Moderate to severe liver hypofunction and severe kidney hypofunction (less than 30 mL/min of creatinine clearance)
9. Any other subjects who are considered to be ineligible for this study by an investigator

[Inclusion Criteria for Randomization]

1. Clinical signs and symptoms of benign prostatic hyperplasia

   1. Volume of prostate gland (TRUS) > 30 cc *
   2. moderate to severe lower urinary tract symptoms with IPSS ≥ 13
   3. 5-15 mL/sec of maximum flow rate (Qmax) measured when urine volume was at least 125 mL
2. Residual urine volume ≤ 200 mL
3. Patient's partner (Consent should be obtained before visit 4, when necessary.) - Consent to avoid pregnancy by using contraceptive devices or oral contraceptives during the patient's participation in clinical trial and for 90 days after the end of treatment, except if the partner reaches menopause or is surgically sterilized.

(* In case that additional TRUS examination has been performed after screening, a decision should be made based on the latest result.)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score(IPSS) | Week 24
  The amount of change from International Prostate Symptom Score(IPSS )compared to the baseline.
  The measures of the 7 items evaluating symptoms is evaluated from 0 to 5 for each item, the total coverage range is from 0 (no symptoms) to 35 (most severe symptoms).
  And the quality of life assessment is assessed from 0 (very satisfactory) to 6 (very unsatisfactory).

SECONDARY OUTCOMES:
Change in International Prostate Symptom Score(IPSS) | Weeks 4, 8, 12, 16 and 20
  The amount of change from International Prostate Symptom Score(IPSS )compared to the baseline.
  The measures of the 7 items evaluating symptoms is evaluated from 0 to 5 for each item, the total coverage range is from 0 (no symptoms) to 35 (most severe symptoms).
  And the quality of life assessment is assessed from 0 (very satisfactory) to 6 (very unsatisfactory).
Change in voiding score of International Prostate Symptom Score(IPSS) | Weeks 4, 8, 12, 16, 20 and 24
  The amount of change from voiding score of IPSS compared to the baseline. The voiding score is measured as the sum of the evaluation scores of items 1, 3, 5 and 6 of the seven symptom scores of the IPSS.
Change in Prostatic Volume(PV) | Weeks 12 and 24
  The amount of change from Prostatic Volume(PV) compared to the baseline.
Change in Maximum(peak) Urinary Flow Rate | Weeks 12 and 24
  The amount of change from Maximum(peak) Urinary Flow Rate compared to the baseline
Change in Prostate-specific Antigen (PSA) | Weeks 12 and 24
  The amount of change from Prostate-specific Antigen (PSA) compared to the baseline
Change in Residual Urine Volume | Weeks 12 and 24
  The amount of change from Residual Urine Volume compared to the baseline
Change in Hormones (Testosterone, DHT) | Weeks 4, 8, 12, 16, 20 and 24
  The amount of change from Hormones (Testosterone, DHT) compared to the baseline
Change in International Index of Erectile Function (IIEF) | Weeks 4, 8, 12, 16, 20 and 24
  The amount of change from International Index of Erectile Function (IIEF) compared to the baseline
rate of incidence of Acute urinary tract(AUR) | Every 2 weeks After screening visit up to 24 week
  The rate of incidence of Acute urinary tract(AUR), meaning clinical progression of prostate hypertrophy
Ratio of prostate surgery and minimally invasive (non-surgical) procedure | Every 2 weeks After screening visit up to 24 week
  The ratio of prostate surgery and minimally invasive (non-surgical) procedure, meaning clinical progression of prostate hypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Seop Lee, Study Chair — Department of Urology, Dongguk University Gyeongju Hospital
Locations (23):
- South Korea (23):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Dongguk University Gyeongju Hospital, Gyeongju, Gyeongsangbuk-do
  - Hallym University Medical Center, Anyang
  - Inje University Busan Paik Hospital, Busan
  - Samsung Changwon Medical Center, Changwon
  - Soonchunhyang University Hospital, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Dongguk University Ilsan Hospital, Ilsan
  - Jeonbuk National University Hospital, Jeonju
  - Chungbuk National University Hospital, Jungbuk
  - Chonnam National University Hospital, Jungnam
  - Asan Medical Center, Seoul
  - Chung-ang University Hospital, Seoul
  - Eulji General Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No